CLINICAL TRIAL: NCT01978873
Title: Randomized Phase III Trial Comparing Cabazitaxel Combination Hormone Therapy to Hormone Therapy Alone in Metastatic Prostate Cancer or High Risk Disease
Brief Title: Efficacy Study Evaluating Chemotherapy in Prostate Cancer
Acronym: SensiCab
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Ove Andrén, MD, Associated professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0030-78-10; 2011-003078-10 (EudraCT Number)
Record Dates: First submitted 2013-02-14; First posted 2013-11-08 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: (Experimental): * Cabazitaxel 25 mg / m² / day on day 1 every 3 weeks continued if the patient has stable disease or responding to up to 10 cycles. Cabazitaxel will be administered in combination with oral prednisone or prednisolone (Prednisolon 10mg 1x1)
  * Hormones will be initiated in conjunction with the last cycle of chemotherapy. Consists of the administration of a luteinizing hormone-releasing hormone (LHRH) agonist + antiandrogens for 30 days OR surgical castration OR complete androgen blockade (CAB) by LHRH agonist + antiandrogen device. G-CSF treatment according to ASCO guidelines is recommended.
  Interventions: Drug: Cabazitaxel + Androgen deprivation therapy
- Arm B: (Active Comparator): -Hormone: LHRH agonist antiandrogens for 30 days + OR surgical castration OR CAB complete androgen blockade by LHRH agonist + antiandrogen device.
  Interventions: Drug: Androgen deprivation therapy

INTERVENTIONS:
Drug: Cabazitaxel + Androgen deprivation therapy — Cabazitaxel + LHRH agonist + antiandrogens for 30 days OR surgical castration OR complete androgen blockade (CAB) by LHRH agonist + antiandrogen device.
  Other Names: Jevtana-Leuporelin
  Arms: Arm A:
Drug: Androgen deprivation therapy — LHRH agonist + antiandrogens for 30 days OR surgical castration OR complete androgen blockade (CAB) by LHRH agonist + antiandrogen device.
  Other Names: Leuporelin
  Arms: Arm B:

SUMMARY:
This clinical trial is designed on the basis of an unmet clinical need, as well as other factors including: 1) the ability to identify subjects at high risk of dying early from their disease, 2) the fact that hormonal therapy has already been shown to improve survival when applied early in the natural history, 3) the availability of chemotherapy such as cabazitaxel that can improve survival in subjects with advanced disease and 4) that chemotherapy (docetaxel) given concomitant with hormone treatment has proven to prolong time to progression.

It is the investigators hypothesis that a more appropriate group of patients who may benefit from the curative potential of systemic chemo-hormonal modality is that with minimal, but detectable disease who have a high probability of developing metastatic disease, clinical symptoms and eventually death from prostate cancer in a defined time frame. The investigators hypothesize further that the approach is likely to be more effective at a time of minimal tumour burden, resulting in minimization of the overall burden of therapy and better quality of life while on treatment.

This trial will determine whether any benefit is gained by adding chemotherapy before hormonal therapy to hormonal therapy alone in the population of subjects with metastatic or high risk disease.

DETAILED DESCRIPTION:
This clinical trial is designed on the basis of an unmet clinical need, as well as other factors including: 1) the ability to identify subjects at high risk of dying early from their disease, 2) the fact that hormonal therapy has already been shown to improve survival when applied early in the natural history, 3) the availability of chemotherapy such as cabazitaxel that can improve survival in subjects with advanced disease and 4) that chemotherapy (docetaxel) given concomitant with hormone treatment has proven to prolong time to progression.

It is the investigators hypothesis that a more appropriate group of patients who may benefit from the curative potential of systemic chemo-hormonal modality is that with minimal, but detectable disease who have a high probability of developing metastatic disease, clinical symptoms and eventually death from prostate cancer in a defined time frame. The investigators hypothesize further that the approach is likely to be more effective at a time of minimal tumour burden, resulting in minimization of the overall burden of therapy and better quality of life while on treatment.

This trial will determine whether any benefit is gained by adding chemotherapy before hormonal therapy to hormonal therapy alone in the population of subjects with metastatic or high risk disease. Two therapeutic approaches will be compared in this two-arm randomized clinical trial. The control Arm A provides hormonal therapy alone. The experimental Arm B involves treatment with hormone therapy + Cabazitaxel 25 mg / m² / day on day 1 every 3 weeks continued if the patient has stable or responding disease up to 10 cycles. For the schematic representation of study design please see Section 7.3.1.

Subjects with primary metastatic or N+ or high risk disease (PSA>100) will be eligible. The primary endpoint of the trial is overall survival.

Based on the yearly number of prostate cancer patients who are diagnosed with metastatic or high risk disease, approximately 1200 men per year (if +15% improvement)are potential candidates for this approach in the Scandinavian countries .

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed prostate adenocarcinoma Metastatic PC (Prostate cancer) with measurable or evaluable disease or High risk PC (PSA > 100) or Node positive disease (N+)
* No prior treatment for prostate cancer (including bisfosfonate)
* Age above 18 years
* ECOG 0- 2
* Estimated survival > 3 months
* WBC 2000 / mm 3, neutrophils ≥1500 / mm 3, platelets 100,000 / mm 3
* Satisfactory liver function: bilirubin, transaminases ≤ 1.5 times the upper limit of normal.
* Satisfactory renal function. Serum creatinine <1.5 x ULN (150 mmol/l). If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance >60 mL/min are accepted in the study. https://www.qxmd.com/calculate-online/nephrology/ckd-epi-egfr
* Patient information and signature of informed consent

Exclusion Criteria:

* Cardiovascular disease (severe symptomatic coronary artery disease, congenital heart failure, class 3 and 4 of the NYHA)
* Severe peripheral neuropathy
* Active infection or other serious underlying pathology that could prevent patients from receiving treatment
* History of cancer within 5 years before inclusion in the study other than basal cell or squamous cell skin cancer adequately treated
* Brain metastases, uncontrolled symptomatic or asymptomatic
* Patient participating in another clinical trial protocol with a molecule during this experimental study or treated four weeks prior to randomization.
* Concurrent or planned treatment with potent inhibitors or inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Appendix A and B)
* Systemic treatment with high dose steroids
* Any severe acute or chronic medical condition which would impair the ability of the patient to participate to the study or interfere with interpretation of study results, or patient unable to comply with the study procedures.
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until date of death from any cause, assessed up to 7 years.

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until progression, assessed up to 3 years.
  Ct and bonescan at three and six months and then at progession. PSA assesments every three moths during the first year and then every six months until progression.
PSA response | From date of randomization up to 7 years.
  Assements every three months during the first year. Then every six months until progression. Then after progression every 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andrén, Ass Prof., Principal Investigator — University Hospital Örebro; Marie Hjelm-Eriksson, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- University Hospital of Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All data from the main study will be made public available after the publication of the study.